CLINICAL TRIAL: NCT01949194
Title: A Phase II Exploratory Study to Identify Biomarkers Predictive of Clinical Response to Regorafenib in Patients With Metastatic Colorectal Cancer Who Have Failed First-line Therapy
Brief Title: Study to Determine the Efficacy of Regorafenib in Metastatic Colorectal Cancer Patients and to Discover Biomarkers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gerald Batist (Other)
Collaborators: Bayer (Industry); Quebec Clinical Research Organization in Cancer (Other)
Responsible Party: Sponsor-Investigator, Gerald Batist, Medical Oncologist, Director Segal Cancer Center, Jewish General Hospital
Organization: Jewish General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QCROC-06
Record Dates: First submitted 2013-09-11; First posted 2013-09-24 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: liver metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regorafenib (Experimental): Single-agent regorafenib
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — The dose of regorafenib given will be 160 mg once a day (od) oral (po), using a 21 days on / 7 days off treatment schedule. This equates to four (4) tablets once a day for three (3) weeks. The patient should take the dose at the same time each day, with a full glass of water, and following a light meal. A "light meal"consists of less than 30% fat and around 300-550 calories.
  Other Names: BAY 73-4506

SUMMARY:
In recent years, anti-angiogenic agents have been incorporated into clinical practice for the treatment of metastatic CRC, leading to improvements in progression-free survival and overall survival. Regorafenib is an oral multi-kinase inhibitor that targets angiogenic and oncogenic kinases. Although structurally similar to another multi-kinase inhibitor, sorafenib, it appears to be pharmacologically more potent and possesses broader antiangiogenic properties.

Both sorafenib and regorafenib target BRAF wild-type and BRAF V600E mutant but the inhibition of p38 MAP kinase is a peculiar characteristic of regorafenib. A Phase I study of regorafenib as a single agent in patients with heavily pretreated CRC showed promising clinical activity with a disease control rate (PR + SD) of 59% in evaluable patients. In the Phase III trial (CORRECT), which was a randomized double-blind, placebo-controlled study comparing either regorafenib plus best supportive care (BSC) or placebo plus BSC, it was shown that regorafenib significantly increased overall survival (OS), progression-free survival (PFS) and disease control rate (DCR), independently of KRAS status. A major interest, given the data presented in the CORRECT trial, is to determine predictive biomarkers to indicate patients likely to benefit, or to be resistant to this anti-angiogenic compound.

This study aims to determine the efficacy of regorafenib as single-agent treatment for the treatment of second-line metastatic colorectal cancer and to identify predictive biomarkers in the actual metastatic tumors to be treated. In the case of metastatic CRC patients, liver lesions are frequently the most common site of metastatic deposit and these lesions can be biopsied to assess putative biomarkers. Patients will be asked to undergo a biopsy of a metastatic lesion prior to treatment, and an optional liver biopsy at the time of relapse. Using several high-throughput discovery platforms, biomarkers will be identified in the metastatic tumor specimens and in blood samples collected throughout the treatment. This will allow us to evaluate putative biomarkers and monitor tumor biomarker dynamics using serial blood collection.

The objectives of this trial are to help identify the patient subgroup most likely to be responsive or resistant to regorafenib, so that future treatment with regorafenib can be directed to the more responsive but as yet identified patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age ≥18 years.
3. Histological documentation of adenocarcinoma of the colon or rectum, with at least one liver metastatic site available for biopsy.
4. Metastatic disease not suitable for upfront curative-intent surgery.
5. Patients must have received one (and no more than one) prior treatment regimen for metastatic CRC.
6. Measurable disease according to RECIST v.1.1.
7. ECOG status ≤1.
8. Life expectancy ≥ 3 months.
9. Women of childbearing potential and men must agree to use adequate contraception since signing of the informed consent form until at least 3 months after the last study drug administration.
10. Adequate bone-marrow, liver, and renal function:

    * Total bilirubin ≤1.5 × ULN
    * ALT and AST ≤5 × ULN (since liver involvement of their cancer)
    * Alkaline phosphatase limit ≤5 × ULN, since liver involvement of their cancer
    * Amylase and lipase ≤1.5 × ULN
    * Serum creatinine ≤1.5 × ULN
    * INR and PTT ≤1.5 × ULN.
    * Platelet count ≥100 x 10^9/L, hemoglobin ≥90 g/L, absolute neutrophil count (ANC) >1.5 x 10^9/L

Exclusion Criteria:

1. Previous treatment with regorafenib.
2. Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years before randomization, EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumours.
3. Extended field radiotherapy within 4 weeks or limited field radiotherapy within 2 weeks prior to registration. Patients must have recovered from all therapy-related toxicities. The site of irradiation should have evidence of progressive disease (new lesions or increase in lesion size) if this is the only site of disease.
4. Major surgical procedure or significant traumatic injury within 28 days before starting the study treatment.
5. Female patients that are pregnant or breast-feeding.
6. Congestive heart failure ≥ Class 2 according to the NYHA.
7. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction less than 6 months before start of study drug
8. Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
9. Uncontrolled hypertension
10. Phaeochromocytoma
11. Pleural effusion or ascites that causes respiratory compromise.
12. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 3 months before starting the study treatment.
13. Ongoing uncontrolled infection > Grade 2 per CTCAE v. 4.0.
14. Known history of HIV infection.
15. Active hepatitis B or C, or chronic hepatitis B or C requiring antiviral therapy.
16. Seizure disorder requiring medication.
17. Any history of or currently known brain metastases (patients with stable brain metastases ≥ 3 months may be eligible for the study).
18. History of organ allograft.
19. Evidence or history of severe bleeding diathesis.
20. Non-healing wound, ulcer, or bone fracture.
21. Renal failure requiring haemodialysis or peritoneal dialysis
22. Dehydration ≥ 2 per CTCAE v. 4.0.
23. Substance abuse or medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
24. Known hypersensitivity to regorafenib, regorafenib class of drugs, or excipients in the formulation.
25. Any illness or medical conditions that are unstable or could jeopardize the safety of the patient in the opinion of the investigator.
26. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
27. Persistent proteinuria ≥ Grade 3 per CTCAE v. 4.0 (i.e. >3.5g/24 hours).
28. Inability to swallow oral medications.
29. Any malabsorption condition.
30. Unresolved toxicity > Grade 1, attributed to any prior therapy/procedure, excluding alopecia and oxaliplatin neurotoxicity ≤ Grade 2, per CTCAE v. 4.0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
A biomarker (in blood or tissue) that may be predictive of level of response to regorafenib | 4 years
  A biopsy from a liver metastasis will be taken at baseline for discovery of biomarkers that correlate with response to regorafenib. Genomic material (DNA and RNA) will be isolated from all biopsies. Those that pass quality control (high quality DNA, RNA and >60% tumor content) will be considered evaluable. Batched analysis will be performed at the end of the study with the evaluable samples for multiplex biomarker discovery. Patient's biomarker status at baseline will be correlated with treatment effect on PFS and response (including response rate and disease control rate) to explore which biological targets may be particularly important in defining the appropriate treatment population for regorafenib.

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 3 years
  Assessment of safety profile of regorafenib in treated patients : report of Adverse Events according to the The NCI's Common Toxicity Criteria version 4.0
Progression free survival (PFS) time | Time from registration to progressive disease (up to 3 years)
  The time from the date of registration until the date of radiological disease progression assessed by RECIST 1.1 or until death due to any cause, even in the absence of radiological progression.
Objective Response Rate (RR) | Up to 3 years
  Determination of the objective response rate (ORR: CR (complete response) +PR (partial response) +SD (stable disease)) of treated patients according to RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Batist, MD, Principal Investigator — Jewish General Hospital; Petr Kavan, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (5):
- Canada (5):
  - The Moncton Hospital (Horizon Health Network), Moncton, New Brunswick
  - Jewish General Hospital, Montreal, Quebec
  - St-Mary's Hospital Centre, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal